CLINICAL TRIAL: NCT02399410
Title: BEV-IP: Perioperative Chemotherapy With Bevacizumab in Patients Undergoing Cytoreduction and Intraperitoneal Chemoperfusion for Colorectal Carcinomatosis
Brief Title: Perioperative Chemotherapy With Bevacizumab for Colorectal Carcinomatosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EC/2014/1042
Record Dates: First submitted 2015-03-09; First posted 2015-03-26 (Estimated); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Colorectal Neoplasms
Keywords: cytoreductive surgery; hipec; perioperative chemotherapy; peritoneal carcinomatosis; bevacizumab; colorectal surgery
MeSH Terms: conditions — Colorectal Neoplasms; Peritoneal Neoplasms | interventions — Bevacizumab; Cytoreduction Surgical Procedures

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- bevacizumab and CRS with oxaliplatin (Experimental): Perioperative chemotherapy plus bevacizumab and CRS with oxaliplatin
  Interventions: Drug: perioperative chemotherapy plus bevacizumab; Procedure: cytoreductive surgery; Drug: Intraperitoneal Oxaliplatin

INTERVENTIONS:
Drug: perioperative chemotherapy plus bevacizumab — preoperative and postoperative combination chemotherapy with bevacizumab
Procedure: cytoreductive surgery — complete or nearly complete removal of synchronous or metachronous peritoneal carcinomatosis from CRC.
Drug: Intraperitoneal Oxaliplatin — Pump-driven intraperitoneal administration of oxaliplatin

SUMMARY:
The Bev-IP trial is designed to assess the feasibility and efficacy of a combined treatment consisting of perioperative combination chemotherapy with the vascular endothelial growth factor A inhibitor bevacizumab and cytoreductive surgery with intraperitoneal oxaliplatin.

ELIGIBILITY:
Inclusion Criteria:

* biopsy proven adenocarcinoma of the colon or rectum and synchronous or metachronous peritoneal carcinomatosis.
* absence of systemic disease, with the exception of small, superficial liver metastases, requiring only minor surgery.
* resectable disease at staging, during laparoscopic evaluation and during exploration for cytoreductive surgery and intraperitoneal chemotherapy.
* complete macroscopic cytoreduction at the time of surgery (CC-0/1)
* good general health status (Karnofsky index > 70%)
* expected life expectancy more than 6 months
* no other malignancy than disease under study
* serum creatinine < 1.5 mg/dl or a calculated GFR ≥ 60 mL/min/1.73 m
* serum total bilirubin < 1.5 mg/dl
* platelet count > 100,000/ml
* hemoglobin > 9g/dl
* neutrophil granulocytes > 1,500/ml
* International Normalized Ration (INR) 2 or < 2
* Absence of alcohol and/or drug abuse
* No inclusion in other clinical trials interfering with the study protocol
* No concurrent chronic systemic immune therapy, chemotherapy, or hormone therapy not indicated in the study protocol
* Absence of heart failure (NYHA 2 or > 2) or significant coronary artery disease
* No pregnancy or breast feeding
* Adequate contraception in fertile patients

Exclusion Criteria:

* No written informed consent
* tumour in the presence of obstruction
* evidence of extra-abdominal disease or extensive liver metastasis
* peritoneal cancer index > 25
* active bacterial, viral or fungal infection
* active gastro-duodenal ulcer
* parenchymal liver disease (any stage cirrhosis)
* uncontrolled diabetes mellitus
* severe obstructive or restrictive respiratory insufficiency
* psychiatric pathology capable of affecting comprehension and judgment faculty
* Known allergy to oxaliplatin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-11-04 (Actual); Primary Completion 2023-11-09 (Actual); Study Completion 2023-11-09 (Actual)

PRIMARY OUTCOMES:
surgical morbidity and mortality | until 3 months after surgery and intraperitoneal chemotherapy
  This will be estimated with the Dindo-Clavien classification

SECONDARY OUTCOMES:
progression free survival | 24 months after finishing the adjuvant chemotherapy
  time interval between date of surgery and disease progression or death
overall survival | 24 months after finishing the adjuvant chemotherapy
  calculated from date of surgery until death
treatment completion rate | day 1 after termination of adjuvant chemotherapy
  percentage of patients receiving all planned courses
chemotherapy-related toxicity | 1 month after termination of the adjuvant chemotherapy
  percentage of patients experiencing chemotherapy-related toxicity will be assessed using the Common Terminology Criteria for Adverse Events (NCI-CTCAE) scoring system
pathological gross response of peritoneal tumour deposits to neoadjuvant combination chemotherapy with bevacizumab | day 1 after termination of the cytoreductive surgery
  will be scored with a 3 level regression scale

CONTACTS AND LOCATIONS:
Overall Officials: Wim P Ceelen, MD,PhD, Principal Investigator — University Hospital, Ghent
Locations (1):
- Ghent University Hospital, Ghent, Belgium

REFERENCES:
- [Background] Herszenyi L, Tulassay Z. Epidemiology of gastrointestinal and liver tumors. Eur Rev Med Pharmacol Sci. 2010 Apr;14(4):249-58. PMID 20496531
- [Background] Peeters M, Price T. Biologic therapies in the metastatic colorectal cancer treatment continuum--applying current evidence to clinical practice. Cancer Treat Rev. 2012 Aug;38(5):397-406. doi: 10.1016/j.ctrv.2011.08.002. Epub 2011 Sep 6. PMID 21899955
- [Background] Klaver YL, Simkens LH, Lemmens VE, Koopman M, Teerenstra S, Bleichrodt RP, de Hingh IH, Punt CJ. Outcomes of colorectal cancer patients with peritoneal carcinomatosis treated with chemotherapy with and without targeted therapy. Eur J Surg Oncol. 2012 Jul;38(7):617-23. doi: 10.1016/j.ejso.2012.03.008. Epub 2012 May 8. PMID 22572106
- [Background] Koppe MJ, Boerman OC, Oyen WJ, Bleichrodt RP. Peritoneal carcinomatosis of colorectal origin: incidence and current treatment strategies. Ann Surg. 2006 Feb;243(2):212-22. doi: 10.1097/01.sla.0000197702.46394.16. PMID 16432354
- [Background] Segelman J, Granath F, Holm T, Machado M, Mahteme H, Martling A. Incidence, prevalence and risk factors for peritoneal carcinomatosis from colorectal cancer. Br J Surg. 2012 May;99(5):699-705. doi: 10.1002/bjs.8679. Epub 2012 Jan 27. PMID 22287157
- [Background] Lemmens VE, Klaver YL, Verwaal VJ, Rutten HJ, Coebergh JW, de Hingh IH. Predictors and survival of synchronous peritoneal carcinomatosis of colorectal origin: a population-based study. Int J Cancer. 2011 Jun 1;128(11):2717-25. doi: 10.1002/ijc.25596. Epub 2010 Oct 13. PMID 20715167
- [Background] Tran B, Kopetz S, Tie J, Gibbs P, Jiang ZQ, Lieu CH, Agarwal A, Maru DM, Sieber O, Desai J. Impact of BRAF mutation and microsatellite instability on the pattern of metastatic spread and prognosis in metastatic colorectal cancer. Cancer. 2011 Oct 15;117(20):4623-32. doi: 10.1002/cncr.26086. Epub 2011 Mar 31. PMID 21456008
- [Background] Sadeghi B, Arvieux C, Glehen O, Beaujard AC, Rivoire M, Baulieux J, Fontaumard E, Brachet A, Caillot JL, Faure JL, Porcheron J, Peix JL, Francois Y, Vignal J, Gilly FN. Peritoneal carcinomatosis from non-gynecologic malignancies: results of the EVOCAPE 1 multicentric prospective study. Cancer. 2000 Jan 15;88(2):358-63. doi: 10.1002/(sici)1097-0142(20000115)88:23.0.co;2-o. PMID 10640968
- [Background] Pelz JO, Chua TC, Esquivel J, Stojadinovic A, Doerfer J, Morris DL, Maeder U, Germer CT, Kerscher AG. Evaluation of best supportive care and systemic chemotherapy as treatment stratified according to the retrospective peritoneal surface disease severity score (PSDSS) for peritoneal carcinomatosis of colorectal origin. BMC Cancer. 2010 Dec 22;10:689. doi: 10.1186/1471-2407-10-689. PMID 21176206
- [Background] Franko J, Shi Q, Goldman CD, Pockaj BA, Nelson GD, Goldberg RM, Pitot HC, Grothey A, Alberts SR, Sargent DJ. Treatment of colorectal peritoneal carcinomatosis with systemic chemotherapy: a pooled analysis of north central cancer treatment group phase III trials N9741 and N9841. J Clin Oncol. 2012 Jan 20;30(3):263-7. doi: 10.1200/JCO.2011.37.1039. Epub 2011 Dec 12. PMID 22162570
- [Background] Euler J, Priesching A, Wenzl J, Sauermann G, Klockler K, Kretschmer G. [Hyperthermic peritoneal perfusion in ascites tumours in rats (author's transl)]. Wien Klin Wochenschr. 1974 Apr 19;86(8):220-5. No abstract available. German. PMID 4822331
- [Background] Spratt JS, Adcock RA, Muskovin M, Sherrill W, McKeown J. Clinical delivery system for intraperitoneal hyperthermic chemotherapy. Cancer Res. 1980 Feb;40(2):256-60. PMID 6766084
- [Background] Hildebrandt B, Wust P, Ahlers O, Dieing A, Sreenivasa G, Kerner T, Felix R, Riess H. The cellular and molecular basis of hyperthermia. Crit Rev Oncol Hematol. 2002 Jul;43(1):33-56. doi: 10.1016/s1040-8428(01)00179-2. PMID 12098606
- [Background] Raaphorst GP, Yang DP. The evaluation of thermal cisplatin sensitization in normal and XP human cells using mild hyperthermia at 40 and 41 degrees C. Anticancer Res. 2005 Jul-Aug;25(4):2649-53. PMID 16080507
- [Background] Los G, Sminia P, Wondergem J, Mutsaers PH, Havemen J, ten Bokkel Huinink D, Smals O, Gonzalez-Gonzalez D, McVie JG. Optimisation of intraperitoneal cisplatin therapy with regional hyperthermia in rats. Eur J Cancer. 1991;27(4):472-7. doi: 10.1016/0277-5379(91)90389-u. PMID 1827723
- [Background] Verwaal VJ, van Ruth S, de Bree E, van Sloothen GW, van Tinteren H, Boot H, Zoetmulder FA. Randomized trial of cytoreduction and hyperthermic intraperitoneal chemotherapy versus systemic chemotherapy and palliative surgery in patients with peritoneal carcinomatosis of colorectal cancer. J Clin Oncol. 2003 Oct 15;21(20):3737-43. doi: 10.1200/JCO.2003.04.187. PMID 14551293
- [Background] Verwaal VJ, Bruin S, Boot H, van Slooten G, van Tinteren H. 8-year follow-up of randomized trial: cytoreduction and hyperthermic intraperitoneal chemotherapy versus systemic chemotherapy in patients with peritoneal carcinomatosis of colorectal cancer. Ann Surg Oncol. 2008 Sep;15(9):2426-32. doi: 10.1245/s10434-008-9966-2. Epub 2008 Jun 3. PMID 18521686
- [Background] Glehen O, Kwiatkowski F, Sugarbaker PH, Elias D, Levine EA, De Simone M, Barone R, Yonemura Y, Cavaliere F, Quenet F, Gutman M, Tentes AA, Lorimier G, Bernard JL, Bereder JM, Porcheron J, Gomez-Portilla A, Shen P, Deraco M, Rat P. Cytoreductive surgery combined with perioperative intraperitoneal chemotherapy for the management of peritoneal carcinomatosis from colorectal cancer: a multi-institutional study. J Clin Oncol. 2004 Aug 15;22(16):3284-92. doi: 10.1200/JCO.2004.10.012. PMID 15310771
- [Background] Yan TD, Black D, Savady R, Sugarbaker PH. Systematic review on the efficacy of cytoreductive surgery combined with perioperative intraperitoneal chemotherapy for peritoneal carcinomatosis from colorectal carcinoma. J Clin Oncol. 2006 Aug 20;24(24):4011-9. doi: 10.1200/JCO.2006.07.1142. PMID 16921055
- [Background] Hompes D, D'Hoore A, Van Cutsem E, Fieuws S, Ceelen W, Peeters M, Van der Speeten K, Bertrand C, Legendre H, Kerger J. The treatment of peritoneal carcinomatosis of colorectal cancer with complete cytoreductive surgery and hyperthermic intraperitoneal peroperative chemotherapy (HIPEC) with oxaliplatin: a Belgian multicentre prospective phase II clinical study. Ann Surg Oncol. 2012 Jul;19(7):2186-94. doi: 10.1245/s10434-012-2264-z. Epub 2012 Mar 7. PMID 22395983
- [Background] Cavaliere F, De Simone M, Virzi S, Deraco M, Rossi CR, Garofalo A, Di Filippo F, Giannarelli D, Vaira M, Valle M, Pilati P, Perri P, La Pinta M, Monsellato I, Guadagni F. Prognostic factors and oncologic outcome in 146 patients with colorectal peritoneal carcinomatosis treated with cytoreductive surgery combined with hyperthermic intraperitoneal chemotherapy: Italian multicenter study S.I.T.I.L.O. Eur J Surg Oncol. 2011 Feb;37(2):148-54. doi: 10.1016/j.ejso.2010.10.014. Epub 2010 Nov 18. PMID 21093205
- [Background] Elias D, Lefevre JH, Chevalier J, Brouquet A, Marchal F, Classe JM, Ferron G, Guilloit JM, Meeus P, Goere D, Bonastre J. Complete cytoreductive surgery plus intraperitoneal chemohyperthermia with oxaliplatin for peritoneal carcinomatosis of colorectal origin. J Clin Oncol. 2009 Feb 10;27(5):681-5. doi: 10.1200/JCO.2008.19.7160. Epub 2008 Dec 22. PMID 19103728
- [Background] Quenet F, Goere D, Mehta SS, Roca L, Dumont F, Hessissen M, Saint-Aubert B, Elias D. Results of two bi-institutional prospective studies using intraperitoneal oxaliplatin with or without irinotecan during HIPEC after cytoreductive surgery for colorectal carcinomatosis. Ann Surg. 2011 Aug;254(2):294-301. doi: 10.1097/SLA.0b013e3182263933. PMID 21772129
- [Background] Franko J, Ibrahim Z, Gusani NJ, Holtzman MP, Bartlett DL, Zeh HJ 3rd. Cytoreductive surgery and hyperthermic intraperitoneal chemoperfusion versus systemic chemotherapy alone for colorectal peritoneal carcinomatosis. Cancer. 2010 Aug 15;116(16):3756-62. doi: 10.1002/cncr.25116. PMID 20564081
- [Background] Cashin PH, Graf W, Nygren P, Mahteme H. Cytoreductive surgery and intraperitoneal chemotherapy for colorectal peritoneal carcinomatosis: prognosis and treatment of recurrences in a cohort study. Eur J Surg Oncol. 2012 Jun;38(6):509-15. doi: 10.1016/j.ejso.2012.03.001. Epub 2012 Apr 3. PMID 22475555
- [Background] Shen P, Hawksworth J, Lovato J, Loggie BW, Geisinger KR, Fleming RA, Levine EA. Cytoreductive surgery and intraperitoneal hyperthermic chemotherapy with mitomycin C for peritoneal carcinomatosis from nonappendiceal colorectal carcinoma. Ann Surg Oncol. 2004 Feb;11(2):178-86. doi: 10.1245/aso.2004.05.009. PMID 14761921
- [Background] Vaira M, Cioppa T, D'Amico S, de Marco G, D'Alessandro M, Fiorentini G, De Simone M. Treatment of peritoneal carcinomatosis from colonic cancer by cytoreduction, peritonectomy and hyperthermic intraperitoneal chemotherapy (HIPEC). Experience of ten years. In Vivo. 2010 Jan-Feb;24(1):79-84. PMID 20133981
- [Result] Ceelen W, Van Nieuwenhove Y, Putte DV, Pattyn P. Neoadjuvant chemotherapy with bevacizumab may improve outcome after cytoreduction and hyperthermic intraperitoneal chemoperfusion (HIPEC) for colorectal carcinomatosis. Ann Surg Oncol. 2014 Sep;21(9):3023-8. doi: 10.1245/s10434-014-3713-7. Epub 2014 Apr 23. PMID 24756812
- [Result] Tamsma JT, Keizer HJ, Meinders AE. Pathogenesis of malignant ascites: Starling's law of capillary hemodynamics revisited. Ann Oncol. 2001 Oct;12(10):1353-7. doi: 10.1023/a:1012504904713. PMID 11762804
- [Result] Welch S, Spithoff K, Rumble RB, Maroun J; Gastrointestinal Cancer Disease Site Group. Bevacizumab combined with chemotherapy for patients with advanced colorectal cancer: a systematic review. Ann Oncol. 2010 Jun;21(6):1152-1162. doi: 10.1093/annonc/mdp533. Epub 2009 Nov 25. PMID 19942597
- [Result] Olsen MW, Ley CD, Junker N, Hansen AJ, Lund EL, Kristjansen PE. Angiopoietin-4 inhibits angiogenesis and reduces interstitial fluid pressure. Neoplasia. 2006 May;8(5):364-72. doi: 10.1593/neo.06127. PMID 16790085
- [Result] Nakahara T, Norberg SM, Shalinsky DR, Hu-Lowe DD, McDonald DM. Effect of inhibition of vascular endothelial growth factor signaling on distribution of extravasated antibodies in tumors. Cancer Res. 2006 Feb 1;66(3):1434-45. doi: 10.1158/0008-5472.CAN-05-0923. PMID 16452199
- [Result] Willett CG, Boucher Y, di Tomaso E, Duda DG, Munn LL, Tong RT, Chung DC, Sahani DV, Kalva SP, Kozin SV, Mino M, Cohen KS, Scadden DT, Hartford AC, Fischman AJ, Clark JW, Ryan DP, Zhu AX, Blaszkowsky LS, Chen HX, Shellito PC, Lauwers GY, Jain RK. Direct evidence that the VEGF-specific antibody bevacizumab has antivascular effects in human rectal cancer. Nat Med. 2004 Feb;10(2):145-7. doi: 10.1038/nm988. Epub 2004 Jan 25. PMID 14745444
- [Result] Kobold S, Hegewisch-Becker S, Oechsle K, Jordan K, Bokemeyer C, Atanackovic D. Intraperitoneal VEGF inhibition using bevacizumab: a potential approach for the symptomatic treatment of malignant ascites? Oncologist. 2009 Dec;14(12):1242-51. doi: 10.1634/theoncologist.2009-0109. Epub 2009 Dec 11. PMID 20008305
- [Derived] Willaert W, Van Der Speeten K, Liberale G, Ceelen W. BEV-IP: Perioperative chemotherapy with bevacizumab in patients undergoing cytoreduction and intraperitoneal chemoperfusion for colorectal carcinomatosis. BMC Cancer. 2015 Dec 16;15:980. doi: 10.1186/s12885-015-1954-x. PMID 26673788